CLINICAL TRIAL: NCT01749878
Title: Study to Assess the Safety and Tolerability of Single Doses of REGN1500
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R1500-HV-1214
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: Cohorts 1 through 6 (Experimental): Group A:
  Cohorts 1 through 3 will receive REGN1500 subcutaneous (SC) or placebo Cohorts 4 through 6 will receive REGN1500 intravenous (IV) or placebo
  Interventions: Drug: REGN1500; Drug: placebo
- Group B (Experimental): Group B will receive REGN1500 IV or placebo
  Interventions: Drug: REGN1500; Drug: placebo
- Group C: Cohorts 1 and 2 (Experimental): Group C:
  Cohort 1 will receive REGN1500 SC or placebo Cohort 2 will receive REGN1500 IV or placebo
  Interventions: Drug: REGN1500; Drug: placebo

INTERVENTIONS:
Drug: REGN1500
Drug: placebo

SUMMARY:
Phase 1, first-in-human, randomized, ascending single-dose, placebo-controlled, double-blind study of the safety, tolerability, and bioeffect of REGN1500

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index 18.0 to 40.0 kg/m2, inclusive
2. Normal standard 12-lead ECG
3. Willing to refrain from the consumption of alcohol for 24 hours prior to each study visit
4. Willing to consistently maintain his/her usual diet for the duration of the study
5. Willing to refrain from strenuous exercise for the duration of the trial
6. Willing and able to comply with clinic visits and study-related procedures
7. Provide signed informed consent
8. For sexually active men and women, willingness to utilize adequate contraception and not have their partner[s] become pregnant during the full duration of the study.

Exclusion Criteria:

1. Any clinically significant abnormalities observed during the screening visit
2. History of drug or alcohol abuse within 1 year of screening
3. Receipt of another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit.
4. Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that may adversely affect the subjects participation in this study
5. Known history of human immunodeficiency virus (HIV) antibody; and/or positive hepatitis B surface antigen (HBsAg), and/or positive hepatitis C antibody (HCV) at the screening visit
6. Hospitalization for any reason within 60 days of screening
7. History or presence of malignancy within 5 years prior to the screening visit (other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, and/or localized carcinoma in situ of the cervix
8. Any medical or psychiatric condition which, in the opinion of the investigator, would place the subject at risk, interfere with participation in the study or interfere with the interpretation of the study results
9. Any subject who is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved in the conduct of the protocol, or family member of staff involved in the conduct of the protocol
10. Pregnant or breast-feeding women

(The inclusion/ exclusion criteria provided above are not intended to contain all considerations relevant to a patient's potential participation in this clinical trial).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety | Day 1 to Day 106/126
  The primary endpoint in the study is the incidence and severity of treatment-emergent adverse events (TEAEs) through day 106/126 in participants treated with REGN1500.

SECONDARY OUTCOMES:
Serum concentration of REGN1500 | Day 1 to Day 106/126
  Serum concentration of REGN1500 over time (summary statistics and PK parameters)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Philadelphia, Pennsylvania
  - Dallas, Texas

REFERENCES:
- [Derived] Ahmad Z, Banerjee P, Hamon S, Chan KC, Bouzelmat A, Sasiela WJ, Pordy R, Mellis S, Dansky H, Gipe DA, Dunbar RL. Inhibition of Angiopoietin-Like Protein 3 With a Monoclonal Antibody Reduces Triglycerides in Hypertriglyceridemia. Circulation. 2019 Aug 6;140(6):470-486. doi: 10.1161/CIRCULATIONAHA.118.039107. Epub 2019 Jun 27. PMID 31242752
- [Derived] Dewey FE, Gusarova V, Dunbar RL, O'Dushlaine C, Schurmann C, Gottesman O, McCarthy S, Van Hout CV, Bruse S, Dansky HM, Leader JB, Murray MF, Ritchie MD, Kirchner HL, Habegger L, Lopez A, Penn J, Zhao A, Shao W, Stahl N, Murphy AJ, Hamon S, Bouzelmat A, Zhang R, Shumel B, Pordy R, Gipe D, Herman GA, Sheu WHH, Lee IT, Liang KW, Guo X, Rotter JI, Chen YI, Kraus WE, Shah SH, Damrauer S, Small A, Rader DJ, Wulff AB, Nordestgaard BG, Tybjaerg-Hansen A, van den Hoek AM, Princen HMG, Ledbetter DH, Carey DJ, Overton JD, Reid JG, Sasiela WJ, Banerjee P, Shuldiner AR, Borecki IB, Teslovich TM, Yancopoulos GD, Mellis SJ, Gromada J, Baras A. Genetic and Pharmacologic Inactivation of ANGPTL3 and Cardiovascular Disease. N Engl J Med. 2017 Jul 20;377(3):211-221. doi: 10.1056/NEJMoa1612790. Epub 2017 May 24. PMID 28538136